CLINICAL TRIAL: NCT03434340
Title: Aromatherapy as Prophylaxis for Prevention of Intrathecal Morphine Induced Nausea and Vomiting in Lower Segment Cesarean Section
Brief Title: Aromatherapy for Prevention of Intrathecal Morphine Induced Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017461
Record Dates: First submitted 2018-01-24; First posted 2018-02-15 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-02

CONDITIONS: Post Operative Nausea and Vomiting
Keywords: peppermint oil; intrathecal morphine; PONV; lower segment cesarean section; dexamethasone; granisetron
MeSH Terms: conditions — Vomiting; Postoperative Nausea and Vomiting | interventions — Granisetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Granisetron & Dexamethasone & Peppermint essential oil (Experimental): Granisetron 1mg and Dexamethasone 4mg administer as intravenous injection once right after delivery of newborn followed by Peppermint essential oil 2 drops on nasal strip applied for 6 hours
  Interventions: Biological: Peppermint essential oil; Drug: Granisetron; Drug: Dexamethasone
- Granisetron & Dexamethasone (Active Comparator): Granisetron 1mg and Dexamethasone 4mg administer as intravenous injection once right after delivery of newborn
  Interventions: Drug: Granisetron; Drug: Dexamethasone

INTERVENTIONS:
Biological: Peppermint essential oil — 2 drops applied on a nasal strip
  Other Names: YoungLiving®, 100% pure Peppermint essential oil
  Arms: Granisetron & Dexamethasone & Peppermint essential oil
Drug: Granisetron — 1mg intravenous injection
Drug: Dexamethasone — 4mg intravenous injection

SUMMARY:
This study evaluates the effect of combining non pharmacological anti emetic prophylaxis, namely peppermint essential oil to granisetron and dexamethasone in patient who receive intrathecal morphine for lower segment cesarean section. Half of the patient will receive nasal strip containing peppermint essential oil in addition to granisetron and dexamethasone while the other half will only receive granisetron and dexamethasone.

DETAILED DESCRIPTION:
It is not uncommon to use different group of anti emetic in order to achieve high successful rate in the prevention of opioid induced nausea and vomiting. This study evaluates the effect of combining non pharmacological and pharmacological method to prevent such condition.

Aromatherapy has been used since many years to treat nausea and vomiting. One of the proposed mechanism is by the activation of olfactory receptor when the molecules of essential oil absorb in the mucus lining olfactory epithelium. The signal is then carried by olfactory sensory neuron to the olfactory bulb which filters and send signal to olfactory cortex as well as limbic system to give the feeling of well being.

Granisetron is a serotonin 3 receptor antagonist prevent or treat nausea and vomiting by competitively blocks the action of serotonin at 5-hydroxytryptamine 3 (5HT3) receptors while the mechanism of action of dexamethasone; which is a glucocorticoids is not fully understood.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I and II.
* Non-smoker.
* BMI =< 40
* Singleton pregnancy

Exclusion Criteria:

* Patient with known allergy to granisetron, dexamethasone, bupivacaine, fentanyl, morphine, paracetamol, celecoxib, ginger oil.
* Patient who has inability to breathe through nose.
* Patient with history of post-operative nausea and vomiting (PONV) or motion sickness

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Severity of nausea and vomiting | 24 hours
  Severity of nausea and vomiting is assessed by direct questioning or spontaneous complaint by patient at three time interval; after institution of spinal anesthesia until prior to being discharged from recovery bay, at 6 hour and 24 hour for 1 day. For nausea, severity is assessed using numerical rating scale (NRS). 0 means no nausea while 10 means worst imaginable nausea. As for vomiting, number of occurrence indicates severity. 1-2 times is considered mild, 3-5 times is moderate and more than 5 times is severe.

CONTACTS AND LOCATIONS:
Overall Officials: Assoc Prof Dr Raha Abdul Rahman, Principal Investigator — Consultant Anaesthesiologist
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ravindran J. Rising caesarean section rates in public hospitals in Malaysia 2006. Med J Malaysia. 2008 Dec;63(5):434-5. PMID 19803313
- [Background] Hines S, Steels E, Chang A, Gibbons K. Aromatherapy for treatment of postoperative nausea and vomiting. Cochrane Database Syst Rev. 2012 Apr 18;(4):CD007598. doi: 10.1002/14651858.CD007598.pub2. PMID 22513952
- [Background] Stoicea N, Gan TJ, Joseph N, Uribe A, Pandya J, Dalal R, Bergese SD. Alternative Therapies for the Prevention of Postoperative Nausea and Vomiting. Front Med (Lausanne). 2015 Dec 16;2:87. doi: 10.3389/fmed.2015.00087. eCollection 2015. PMID 26734609
- [Background] Carvalho FA, Tenorio SB. Comparative study between doses of intrathecal morphine for analgesia after caesarean. Braz J Anesthesiol. 2013 Nov-Dec;63(6):492-9. doi: 10.1016/j.bjane.2013.01.001. Epub 2013 Dec 5. PMID 24565347
- [Background] Allen TK, Jones CA, Habib AS. Dexamethasone for the prophylaxis of postoperative nausea and vomiting associated with neuraxial morphine administration: a systematic review and meta-analysis. Anesth Analg. 2012 Apr;114(4):813-22. doi: 10.1213/ANE.0b013e318247f628. Epub 2012 Feb 17. PMID 22344239
- [Background] Gehling M, Tryba M. Risks and side-effects of intrathecal morphine combined with spinal anaesthesia: a meta-analysis. Anaesthesia. 2009 Jun;64(6):643-51. doi: 10.1111/j.1365-2044.2008.05817.x. PMID 19462494
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162
- [Background] Shanazi M, Farshbaf Khalili A, Kamalifard M, Asghari Jafarabadi M, Masoudin K, Esmaeli F. Comparison of the Effects of Lanolin, Peppermint, and Dexpanthenol Creams on Treatment of Traumatic Nipples in Breastfeeding Mothers. J Caring Sci. 2015 Dec 1;4(4):297-307. doi: 10.15171/jcs.2015.030. eCollection 2015 Dec. PMID 26744729
- [Background] Cooke B, Ernst E. Aromatherapy: a systematic review. Br J Gen Pract. 2000 Jun;50(455):493-6. PMID 10962794
- [Derived] Griffiths JD, Gyte GM, Popham PA, Williams K, Paranjothy S, Broughton HK, Brown HC, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2021 May 18;5(5):CD007579. doi: 10.1002/14651858.CD007579.pub3. PMID 34002866